CLINICAL TRIAL: NCT00957216
Title: Safety and Tolerability of Coenzyme Q10 in Adult-Onset Sporadic Spinocerebellar Ataxia
Brief Title: Coenzyme Q10 in Adult-Onset Ataxia
Acronym: CoQATAX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 08-129; 08-SAOA-001
Record Dates: First submitted 2009-06-22; First posted 2009-08-12 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2010-04

CONDITIONS: Sporadic Ataxia
Keywords: adult onset ataxia
MeSH Terms: interventions — Sugars; coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo (sugar pill)
- Coenzyme Q10 (Active Comparator): The CoQ10 arm will be compared with the placebo arm to determine if high-dose CoQ10 is safe and well tolerated in subjects with sporadic adult-onset spinocerebellar ataxias
  Interventions: Drug: Coenzyme Q10

INTERVENTIONS:
Drug: Placebo (sugar pill) — placebo: 2 wafers 4 times a day
  Arms: sugar pill
Drug: Coenzyme Q10 — 300mg wafers; 2 wafers 4 times a day
  Other Names: CoQ10
  Arms: Coenzyme Q10

SUMMARY:
This is a Physician-sponsored pilot study, whose purpose it is determine if high-dose oral Coenzyme Q10 (CoQ10) is safe and tolerated in patients with sporadic forms of adult-onset spinocerebellar ataxias (SAOA), a group of degenerative neurological disorders affecting the cerebellum and pathways to and from the cerebellum, with or without additional central nervous system (CNS) manifestations, in the absence of family history of degenerative ataxias.

DETAILED DESCRIPTION:
This is a Physician-sponsored pilot study, whose purpose it is determine if high-dose oral Coenzyme Q10 (CoQ10) is safe and tolerated in patients with sporadic forms of adult-onset spinocerebellar ataxias (SAOA), a group of degenerative neurological disorders affecting the cerebellum and pathways to and from the cerebellum, with or without additional central nervous system (CNS) manifestations, in the absence of family history of degenerative ataxias.

CoQ10 is an essential cofactor of the electron transport chain and is a potent free radical scavenger in lipid and mitochondrial membranes. CoQ10 has shown efficacy in treatment of Parkinson's disease patients, and a Huntington's disease trial gave a trend of slowing down disease progression (CARE-HD). A small trial of CoQ10 in patients with Friedreich's ataxia suggested potential beneficial effects on ventricular thickness. CoQ10 is being tested on ALS patients and is considered to be potentially useful for treatment of Alzheimer's disease. Thus, CoQ10 is considered to be a promising therapeutic agent that might slow down the disease progression in a wide variety of neurodegenerative disorders. To date, very high doses of CoQ10 have not been used in patients with ataxia and the safety and tolerability in this group of patients should be established before efficacy trials are launched.

Twenty patients with SAOA will be recruited for a double-blind, randomized, placebo-controlled, multicenter study. Fifteen patients will receive a total of 2400 mg of oral CoQ10 daily, and five patients will receive placebo, for a period or 4 weeks. Cerebellar functions will be measured using a validated rating scale (SARA), an oculomotor examination, and functional measurement of motor function using a 9 hole peg test and timed walk. Safety labs will be collected and a digital movie will be recorded at the beginning (prior to treatment with CoQ10) and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SAOA
2. Age 18 or older
3. Adult onset of ataxia
4. Ambulatory capability (with or without an assisting device)
5. Women with 2 years post menopause or surgical sterility or practicing adequate birth control
6. Stable doses of psychotropic drugs
7. Stable doses of drugs for movement disorders
8. Ability to give informed consent
9. Ability to comply with trial procedures
10. Able to take oral medication
11. No active and significant systemic disease (cardiac, pulmonary, hepatic, renal disease or cancer) that is not under adequate medical control
12. Women with child-bearing potential who have a negative urine pregnancy test and practice adequate contraception during the study

Exclusion Criteria:

1. A history or known sensitivity of intolerability to Coenzyme Q10
2. Diagnosis of secondary (non-degenerative) ataxia
3. Family history of degenerative ataxia
4. Diagnosis of childhood-onset ataxia
5. DNA diagnosis of inherited ataxia in the absence of family history
6. Other investigational agent within 30 days of screening
7. Ingestion of Coenzyme Q10 within 120 days of the baseline visit
8. Diagnosis of ongoing malignancy
9. Women who are pregnant or lactating or who have child bearing potential and not using effective birth control
10. Uncontrolled hypertension
11. Symptomatic orthostatic hypotension
12. Uncontrolled diabetes mellitus
13. Untreated thyroid disease
14. Major psychiatric disease within 12 months of screening
15. History of non-compliance with other therapies
16. Drug or alcohol abuse within 12 months of screening
17. Other condition or therapy that may prevent participation in the opinion of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Measure cerebellar functions by a validated scale (SARA) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sankarasubramoney H Subramony, MD, Principal Investigator — University of Texas Medical Branch, Galveston
Locations (1):
- The Universtity of Texas, Galveston, Galveston, Texas, United States